CLINICAL TRIAL: NCT06025734
Title: Effectiveness of Transcutaneous Tibial Nerve Stimulation in Pediatric Patients With Neurogenic Bladder Secondary to Spina Bifida
Brief Title: Transcutaneous Tibial Nerve Stimulation (TTNS) Treatment in Spina Bifida Pediatric Patients With Neurogenic Bladder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Richard Adams, Professor, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STU-2023-0178
Record Dates: First submitted 2023-08-22; First posted 2023-09-06 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Spina Bifida
Keywords: Pediatrics; Neurogenic bladder; TTNS
MeSH Terms: conditions — Spinal Dysraphism; Urinary Bladder, Neurogenic | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- TTNS Treatment Arm (Experimental): Treatments Patient will complete 6 weeks of 30 minute treatment sessions (these can be done at home after the first teaching session) During treatments, patient may experience a tingling sensation in the foot/ankle. Patient may have discomfort in the area when first adjusting to the correct amount of stimulation for patient.
  Patient will have a visit with your doctor after 6 weeks of treatment at Scottish Rite. If patient have a good response to the treatments, they may be extended for another 6 weeks.
  After treatments Bladder diary (completed at home, on paper over a 3-day period, recording catheterization volumes and amount of leakage by weighing pads/diapers) Complete questionnaires on paper (about 10 minutes) Complete urodynamic testing at Children's Medical Center (approximately 45-60 minutes).
  Interventions: Device: Transcutaneous Tibial Nerve Stimulation (TTNS) treatment

INTERVENTIONS:
Device: Transcutaneous Tibial Nerve Stimulation (TTNS) treatment — Spina Bifida pediatric patients with neurogenic bladder will be in Transcutaneous Tibial Nerve Stimulation (TTNS) treatment. Patient will complete 6 weeks of 30 minute treatment sessions (these can be done at home after the first teaching session)

SUMMARY:
The purpose of this research study is to determine the effectiveness of a treatment called "transcutaneous tibial nerve stimulation" or "TTNS" in the treatment of urinary leakage for patients with spina bifida. This treatment involves electrical stimulation of a nerve by the ankle. Participants will complete urodynamic testing and questionnaires prior to the treatments. Participants will then complete 6 weekly treatments of TTNS. Participants will learn how to do the treatment in the clinic, and then can complete the treatments at home. For patients with a good response, the treatments may be continued for another 6 weeks, for a total of 6 weeks.

DETAILED DESCRIPTION:
This study is designed to determine the outcomes of spina bifida patients with neurogenic bladder who receive Transcutaneous Tibial Nerve Stimulation (TTNS) treatment.

To identify patients that may receive the most benefit from TTNS treatment.

Patients with neurogenic bladder secondary to spina bifida with low-risk bladders, who are compliant with catheterizing, will see decreased urinary leakage and improved urodynamic parameters when used in combination with TTNS treatment.

Posterior tibial nerve stimulation via percutaneous (PTNS) or transcutaneous (TTNS) approaches have been effective in treating urinary incontinence from overactive bladder (OAB) and voiding dysfunction in adults. While the exact mechanism of action remains under evaluation, it is a standard of care for adults with OAB refractory to behavioral modifications. Studies have shown PTNS to be effective in children with overactive bladder disease and urinary retention secondary to non-neurogenic causes. TTNS has been shown to be effective for OAB symptoms in children compared to sham intervention, and further studies are ongoing. Moreover, it has been demonstrated that TTNS is non-inferior to PTNS in treating OAB in adults. TTNS is appealing due to its less invasive nature compared to PTNS.

Posterior tibial nerve stimulation implementation in the pediatric population is increasing. To date, few studies have evaluated the efficacy of posterior tibial nerve stimulation in children with spina bifida as some believe the spinal dysraphism may disrupt the mechanism of the technique. However, another form of neuromodulation, surgically-implanted sacral neuromodulation (Interstim), has been shown to be effective for urinary and bowel parameters for some patients with neurogenic bladder secondary to spina bifida. The hypothesis in the proposed study is that TTNS may benefit a subset of patients with less severe spina bifida and may be a treatment option in managing their refractory urinary incontinence.

Pre-intervention

If patient is on bladder medication(s) (anticholinergics or beta agonists), they will stop the bladder medication 2-4 weeks (minimum of 2 weeks) before pre-intervention urodynamic study (UDS)

Patient will complete 3 Day Bladder Diary at home prior to intervention (must be done at least 2 weeks after stopping bladder medications)

Patients will be provided scales for measuring diaper/pad weights at home.

At least 2 weeks after stopping bladder medications (if applicable), patient completes UDS (standard, not video) at Children's Medical Center (CMC)

At this visit, patient completes pre-intervention questionnaires (detailed below in Section 7)

Intervention Period

Intervention overview: Patients will complete weekly 30-minute sessions of TTNS. Intervention procedure described below.

The intervention period will start as 6 weeks for all patients, with extension to 12 weeks for patients who meet any of the measures of success as defined below in the "Post-intervention" section

After patient has completed pre-intervention 3 Day Bladder Diary, UDS and questionnaires, they will proceed with TTNS nursing teaching visit and the first TTNS session at Texas Scottish Rite Hospital (TSRH) or Children's Medical Center Dallas (therefore, if they have completed the Bladder Diary prior to their UDS appointment, the TTNS nursing teaching visit can be completed the same day as their UDS appointment)

At the teaching visit, patient/parent will be shown how to perform the TTNS treatment. They will then demonstrate the process of placing the electrodes and starting the treatment. The first 30-minute session will then be done at this visit. If understanding of process is demonstrated, further treatments will be done at home. If not, they will return the following week for further teaching and the second treatment. Nursing visits will be continued until proficiency is demonstrated by the patient/family, as assessed by the nurse conducting the visit.

The patient will be contacted by phone by the research team weekly after their nursing visit when proficiency was demonstrated, in order to answer questions and monitor compliance. Patients will return for additional teaching sessions as needed.

ELIGIBILITY:
Inclusion Criteria:

* Age 8-18
* Patient at TSRH
* Diagnosis of lumbosacral spina bifida (myelomeningocele, meningocele, lipoma of spinal cord, myelocystocele, diastematomyelia, fatty/thickened filum)
* Incontinence refractory to compliant catheterization (compliance with catheterization as assessed by their treating provider)
* Patient able and willing to undergo urodynamic testing without sedation
* No surgical reconstruction with the exception of a single appendicovesicostomy (APV)
* No Botox treatments within 1 year of enrollment
* Patient willing and able to stop bladder medications (anticholinergics or beta agonists) 2 weeks prior to pre-intervention bladder diary, questionnaires and UDS
* Patient lives close enough to TSRH and CMC to be willing to return for UDS, teaching, and clinic visits as detailed above
* Patient/family speak English

Exclusion Criteria:

* Ages <8 or >18
* Diagnosis not listed above
* Patients that have received reconstructive surgeries (i.e. augmentation or bladder neck sling) with the exception for a single APV
* Patient received Botox treatment within 1 year of enrollment
* Patient unable or unwilling to stop bladder medications (anticholinergics or beta agonists)
* Patients with high-risk bladders, as assessed by their treating provider (i.e. poorly compliant bladders with high end-fill pressures)
* Non-English speaking
* Patients who are pregnant
* Patients who are suspected of being pregnant
* Patients who are nursing

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-11-18 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Number of leakage episodes | 12 weeks
  Number of leakage episodes will be measured by 3 Day Bladder Diary

SECONDARY OUTCOMES:
Leak weight | 12 weeks
  Leak weight of the diapers will be measured by wet-diaper weight in grams
Number of pads used | 12 weeks
  Number of pads used will be measured using 3-day bladder diary
Number of diapers used | 12 weeks
  Number of diapers used will be measured using 3-day bladder diary
Quality of Life Assessment in Spina Bifida Score | 12 weeks
  Quality of life (QoL) is measured by QUALAS assessment tool. QUALAS stands for Quality of Life Assessment of spina bifida. There are separate (but largely similar) versions for adults (QUALAS-A), children aged 8-12 (QUALAS-C) and teenagers (QUALAS-T). Each of these have further "domains" (that are scored from 0-100) that are aggregated to report quality of life scores (see below): 2 domains each for QUALAS C and T, and 3 domains for QUALAS-A. Lower scores in C and T indicate better QoL. But in QUALAS A it is mixed (Domain 1 -'Health and Relationships' : Higher scores indicate better QoL; Domain 2- 'Esteem and Sexuality' : Lower scores indicate better QoL ; Domain 3- 'Bowel and Bladder' : Lower scores indicate better QoL)
Self assessment of improvement | 12 weeks
  Improvement will be measured quantitatively in 1-5 range where 1 reflects strong disagreement and 5 strong agreement

CONTACTS AND LOCATIONS:
Overall Officials: Richard Adams, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- Scottish Rite for Children, Dallas, Texas, United States